CLINICAL TRIAL: NCT00001214
Title: Lymphocytapheresis of Patients With Pancytopenia
Brief Title: Collection of Blood From Patients With Pancytopenia
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 860088; 86-H-0088
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Pancytopenia
Keywords: Bone Marrow Failure; Lymphocytapheresis; Pancytopenia; Aplastic Anemia; Hematosuppressive Disease
MeSH Terms: conditions — Pancytopenia; Bone Marrow Failure Disorders; Anemia, Aplastic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients with pancytopenia

SUMMARY:
Aplastic anemia is a condition in which the cells normally found in blood are greatly decreased. The normal levels of white blood cells, red blood cells, and platelets are much lower in patients with aplastic anemia.

Because of these low levels of blood cells, patients with aplastic anemia have a variety of immune system abnormalities. However, low levels of blood cells make it difficult to collect specialized white blood cells (mononuclear cells) for research studies.

This study was designed to collect lymphocytes from patients with low levels of all blood cells (pancytopenia) for use in research. Patients participating in the study will undergo a special procedure known as lymphapheresis. During lymphapheresis blood is taken from the patient in a manner similar to blood donation. The white blood cells are selectively removed by spinning (centrifugation), and the remaining red blood cells and platelets are placed back (re-infused) into the donor s blood stream.

Patients participating in this study will not benefit directly from it. However, cells collected in this study may increase scientific knowledge and improve understanding and treatment for diseases like aplastic anemia.

DETAILED DESCRIPTION:
Patients with aplastic anemia, myelodysplasia, and other marrow failure syndromes have a variety of immunologic abnormalities including lymphocyte phenotypic and lymphokine production dysregulation. Because of their low blood counts, it has been difficult to obtain sufficient peripheral blood mononuclear cells for research studies. Patients agreeing to this protocol will be lymphapheresed the equivalent of one or two units of cells (approximately 1-2 x 10(8) cells), which will be used for research purposes.

ELIGIBILITY:
* INCLUSION CRITERIA:

All patients with aplastic anemia or other bone marrow failure in which we would not expect to obtain 1 X 10(8) mononuclear cells from 100 mls of peripheral blood (i.e. an absolute lymphocyte count approximately less than 2000 per mm(3)).

Age greater than or equal to 18.

EXCLUSION CRITERIA:

Patients unable to comprehend the investigational nature of the procedure.

Patients unable to tolerate a temporary reduction of blood volume the equivalent of one unit of blood.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancytopenia@@@
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 1986-04-30 (Actual); Primary Completion 2009-01-19 (Actual); Study Completion 2020-08-17 (Actual)

PRIMARY OUTCOMES:
Goal was to obtain adequate numbers of cells for laboratory studies from pancytopenic patients in whom simple phlebotomy is inadequate. | 1 day
  To obtain enough cells if phlebotomy inadequate.

CONTACTS AND LOCATIONS:
Overall Officials: Neal S Young, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1986-H-0088.html